CLINICAL TRIAL: NCT05966857
Title: FAPO-X: Assisted Digital Telemonitoring With Wearables in Patients After Cardiovascular Surgery
Acronym: FAPO-X
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Fabio Biscegli Jatene, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 66520122.0.0000.0068
Record Dates: First submitted 2023-07-07; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result

STUDY DESIGN:
Intervention Model Description: This interventional study utilized a parallel assignment model to develop and validate an assisted digital telemonitoring platform for patients with POAF. The telemonitored group received interventions and telemonitoring through the platform, while the control group followed the standard institutional patient journey without any intervention or telemonitoring.
Who Masked: Outcomes Assessor
Masking Description: During the 30-day telemonitoring period in the TLM (Telemonitoring) group, the ECG report evaluator was blinded to the patient's clinical condition and the presence of underlying atrial fibrillation (AF).
  This masking approach was adopted to ensure that the evaluator was not influenced by prior clinical information or knowledge of the presence of AF before analyzing the ECG results provided by the smartwatch. The objective is to ensure impartiality and objectivity in the evaluation of the data obtained during the telemonitoring period.
  By keeping this information hidden from the evaluator, a more unbiased and accurate analysis of the results can be achieved, without the influence of prior knowledge about the patient's clinical condition or the presence of AF. This contributes to ensuring the validity and reliability of the results obtained through smartwatch telemonitoring in the TLM group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CTL) (No Intervention): Patients who underwent standard treatment at the institution without any wearable monitoring.
- Telemonitored Group (TLM) (Experimental): Patients who received telemonitoring with a Samsung Galaxy smartwatch and FAPO SI³ platform, which is integrated with the hospital's electronic medical record system.
  Interventions: Device: Wearable: Smartwatch

INTERVENTIONS:
Device: Wearable: Smartwatch — The SAMSUNGTM Galaxy Watch5 Smartwatch, is a new generation of smartwatches, features an innovative 3-in-1 BioActive sensor, which uses a chip to capture optical and read cardiac electrical current, allowing to carry out high-quality real-time single-lead electrocardiogram. Despite the more compact design, there is no decrease in accuracy. These signals are then processed by the device's algorithms and can be sent to a trained professional for evaluation immediately after the measurement, facilitating the monitoring and diagnosis of arrhythmias.
  Arms: Telemonitored Group (TLM)

SUMMARY:
This study aims to develop a digitally assisted telemonitoring platform using the Samsung TM Galaxy Watch5 smartwatch, validating the applicability of the solution in patients with POAF (Postoperative Atrial Fibrillation), along with the accuracy of the smartwatch in detecting vital signs through optical sensors and possibly identifying irregularities in heart rhythm. The validation of its applicability will be carried out through a clinical trial. This is a randomized observational pilot study resulting from the partnership established in the base year of 2022 between InCor and Samsung.

The sample consisted of 108 outpatient patients with cardiac diseases who underwent cardiac surgery and were selected during the preoperative consultation. Subsequently, the patients were randomized (1:1) into the intervention group (teleassisted group) or the control group (standard institution follow-up).

The sample size was proposed by the contracting party as this is a pilot study to assess whether the implementation of a technological solution assists in monitoring and predicting the risk of surgical patients in the postoperative phase, as well as the accuracy of the Samsung TM Galaxy Watch5 smartwatch in a sample with POAF.

DETAILED DESCRIPTION:
This interventional study was conducted exclusively at the Heart Institute of the Clinics Hospital of the Medical School of the University of São Paulo (InCor - HCFMUSP). It was a single-center study divided into six phases.

The first phase involved outpatient preoperative care, where patients underwent a comprehensive anamnesis during the preoperative consultation and were informed about the study. In the second phase, patients were hospitalized and provided with the Informed Consent Form (ICF) if they met the inclusion criteria. Demographic data were collected during this phase.

During the surgical phase (third phase), intraoperative data were collected after cardiac surgery. The fourth phase focused on postoperative care, where patients were evaluated, and health measures such as blood pressure (BP), heart rate (HR), electrocardiogram (ECG), and peripheral oxygen saturation (SpO2) were collected using the SAMSUNGTM Galaxy Watch5 smartwatch and reference devices.

After discharge, the fifth phase involved a 30-day telemonitoring period, where patients were remotely monitored using the smartwatch. Health data, including BP, HR, ECG, and SpO2, were collected three times a day during this phase. The medical team provided clinical interventions when alerts were received via the "FAPO SI³" platform.

In the final phase, patients returned for an outpatient visit at InCor, where health measures were collected again using the smartwatch and reference devices. Additionally, a World Health Organization Quality of Life (WHOQOL) questionnaire was administered to assess patients' quality of life. ECG reports issued by the smartwatch were also reviewed.

The control group consisted of patients with heart disease who underwent surgical procedures and received standard outpatient and post-surgical follow-up according to institutional routines and protocols.

Overall, the study aimed to develop and validate an assisted digital telemonitoring platform for patients with postoperative atrial fibrillation (POAF). The telemonitored group used the SAMSUNGTM Galaxy Watch5 smartwatch for remote monitoring, while the control group followed standard care protocols.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years;
* Parameters for surgical indication, in the presence of heart disease (mitral or aortic valve disease, coronary artery disease or aortic disease);
* Agree to adhere to the study's procedures and requirements;
* Be able to consent to their participation in writing;

Exclusion Criteria:

* Not having undergone cardiac surgery;
* Presence of post-surgical complications with prolonged hospital stay for more than 14 days from surgery date;
* Presence of a Peripherally Inserted Central Catheter (PICC) or limb preservation and cardiac pacemaker in case of impediment to acquisition of the ECG (smartwatch);
* Patients with arteriovenous fistula;
* Presence of skin pathology or skin diseases such as vitiligo, lupus and atopic dermatitis, as well as tattoos in the wrist region, which may interfere with the reading by the optical sensor;
* Show sensitivity or allergic reactions, to any degree, to the component materials of the wearable device;

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Rehospitalization rate | 30-day
  Frequency (n, %)
Scheduled consultations | 30-day
  Frequency (n, %)
Extra occurences | 30-day
  Frequency (n, %)

SECONDARY OUTCOMES:
Technological adherence | 30-day
  Frequency (n, %)
Treatment adherence | 30-day
  Frequency (n, %)
Use of the mobile application by patients | 30-day
  Frequency (n, %)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coracao (Heart Institute), Faculdade de Medicina, Hospital das Clinicas, Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Lippi G, Sanchis-Gomar F, Cervellin G. Global epidemiology of atrial fibrillation: An increasing epidemic and public health challenge. Int J Stroke. 2021 Feb;16(2):217-221. doi: 10.1177/1747493019897870. Epub 2020 Jan 19. PMID 31955707
- [Result] Albini A, Malavasi VL, Vitolo M, Imberti JF, Marietta M, Lip GYH, Boriani G. Long-term outcomes of postoperative atrial fibrillation following non cardiac surgery: A systematic review and metanalysis. Eur J Intern Med. 2021 Mar;85:27-33. doi: 10.1016/j.ejim.2020.12.018. Epub 2021 Jan 2. PMID 33402281
- [Result] Lopes LA, Agrawal DK. Post-Operative Atrial Fibrillation: Current Treatments and Etiologies for a Persistent Surgical Complication. J Surg Res (Houst). 2022;5(1):159-172. doi: 10.26502/jsr.10020209. Epub 2022 Mar 28. PMID 35445200
- [Result] Goulden CJ, Hagana A, Ulucay E, Zaman S, Ahmed A, Harky A. Optimising risk factors for atrial fibrillation post-cardiac surgery. Perfusion. 2022 Oct;37(7):675-683. doi: 10.1177/02676591211019319. Epub 2021 May 26. PMID 34034586
- [Result] Phan K, Ha HS, Phan S, Medi C, Thomas SP, Yan TD. New-onset atrial fibrillation following coronary bypass surgery predicts long-term mortality: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2015 Dec;48(6):817-24. doi: 10.1093/ejcts/ezu551. Epub 2015 Jan 18. PMID 25602053
- [Result] Baig MM, GholamHosseini H, Moqeem AA, Mirza F, Linden M. A Systematic Review of Wearable Patient Monitoring Systems - Current Challenges and Opportunities for Clinical Adoption. J Med Syst. 2017 Jul;41(7):115. doi: 10.1007/s10916-017-0760-1. Epub 2017 Jun 19. PMID 28631139
- [Result] Tison GH, Sanchez JM, Ballinger B, Singh A, Olgin JE, Pletcher MJ, Vittinghoff E, Lee ES, Fan SM, Gladstone RA, Mikell C, Sohoni N, Hsieh J, Marcus GM. Passive Detection of Atrial Fibrillation Using a Commercially Available Smartwatch. JAMA Cardiol. 2018 May 1;3(5):409-416. doi: 10.1001/jamacardio.2018.0136. PMID 29562087
- [Result] Chandrasekaran R, Katthula V, Moustakas E. Patterns of Use and Key Predictors for the Use of Wearable Health Care Devices by US Adults: Insights from a National Survey. J Med Internet Res. 2020 Oct 16;22(10):e22443. doi: 10.2196/22443. PMID 33064083
- [Result] Nachman D, Gilan A, Goldstein N, Constantini K, Littman R, Eisenkraft A, Grossman E, Gepner Y. Twenty-Four-Hour Ambulatory Blood Pressure Measurement Using a Novel Noninvasive, Cuffless, Wireless Device. Am J Hypertens. 2021 Nov 20;34(11):1171-1180. doi: 10.1093/ajh/hpab095. PMID 34143867

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT05966857/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT05966857/ICF_001.pdf